CLINICAL TRIAL: NCT05972629
Title: A Phase 1/Phase 2, Open-label, Dose-escalation, and Dose Expansion Study to Evaluate the Safety, Tolerability, and Efficacy of SAR444836, an Adeno-associated Viral Vector-mediated Gene Transfer of Human Phenylalanine Hydroxylase, in Adult Participants With Phenylketonuria
Brief Title: A Phase 1/Phase 2 Open-label Study to Evaluate the Safety, Tolerability, and Efficacy of a Single Intravenous Administration of SAR444836 in Adult Participants With Phenylketonuria
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI17545; U1111-1271-1293 (Registry Identifier: ICTRP); 2022-501200-98 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-06-23; First posted 2023-08-02 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR444836 (Experimental): Participants will receive a single dose of SAR444836 on Day 1
  Interventions: Drug: SAR444836

INTERVENTIONS:
Drug: SAR444836 — Infusion pump, intravenous infusion (IV)

SUMMARY:
This is a single group Phase 1/Phase 2, 1-arm, open-label study with SAR444836, an adeno-associated virus (AAV) vector-mediated gene transfer of human phenylalanine hydroxylase (PAH), for the treatment of adult participants with phenylketonuria (PKU) on a chronic, stable diet. The purpose of the study is to evaluate the safety and efficacy of SAR444836 in reducing phenylalanine (Phe) levels and in the elimination of a Phe restricted diet.

Participants will receive a one-time intravenous (IV) administration of SAR444836.

The study is constituted of 2 separate parts: a dose escalation part, and a dose expansion part where subsequent participants will be administered a safe and effective dose level identified during the dose escalation part. In both study parts, clinical and laboratory assessments will be collected to: a) assess the incidence of adverse events, and b) evaluate the effect of SAR444836 on reductions in blood Phe levels and maintenance of these Phe levels after elimination of a Phe restricted diet.

The study duration will be for a minimum duration of 5 years following SAR444836 administration, for each participant and includes a 6-week screening phase, a 96-week treatment follow-up period after SAR444836 administration, followed by an additional 3 years of long-term safety (and efficacy) monitoring.

There will be a total of 47 study visits. Many study visits may occur as remote visits and be performed by a qualified in-home service provider.

Actual study duration for an individual participant may be longer than 5 years due to the administration of SAR444836 to participants in Stage 1A in a serial fashion, the duration of the screening period, and/or other factors such as delays in scheduling study visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult males, and females of non-childbearing potential, 18-65 years of age at the time of informed consent.
* Participants must have uncontrolled classical PKU due to PAH deficiency (despite Phe-restricted dietary management or Palynziq) in the judgement of the Investigator.
* Two historical plasma Phe values ≥ 600 μmol/L in the preceding 12 months while on Phe restricted diet therapy. Two plasma Phe values ≥ 600 μmol/L drawn at least 72 hours apart during the screening period while on Phe restricted diet therapy in the absence of an acute illness.
* Participant has the ability and willingness to maintain their present diet for the duration of the Post-treatment Follow-up Phase (through Week 96), unless otherwise directed as per protocol
* Body mass index (BMI) ≤ 35 kg/m2
* Willingness to use effective methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Presence of neutralizing antibodies against the AAV SNY001 capsid
* Abnormal liver function laboratory testing evidenced by alanine aminotransferase (ALT)>1.5X upper limit normal (ULN), aspartate transaminase (AST)>1.5X ULN, alkaline phosphatase >1.5X ULN, Total and direct bilirubin >1.5X ULN (bilirubin levels above the laboratory's normal range are acceptable in individuals with a documented history or laboratory evidence of Gilbert's Disease)
* Any significant underlying liver disease or any of the following documented diagnoses, indicative of significant underlying liver disease:

  * Portal hypertension; or
  * Splenomegaly; or
  * Hepatic encephalopathy
* Serum albumin measurement below the lower limit of normal of the laboratory OR AST-to-Platelet Ratio Index > 1.0
* Serum creatinine >1.5X ULN
* Hemoglobin A1c >6.5% or fasting glucose >126 mg/dL
* Screening laboratory testing demonstrating any of the following:

  * HIV; or
  * active or prior hepatitis B virus (HBV) infection defined as positive test for hepatitis B surface antigen (HBsAg) or positive test for hepatitis B core antibody (total HBcAb) or detectable HBV DNA; or
  * active hepatitis C virus (HCV) infection defined as positive test for hepatitis C antibody followed by detectable HCV RNA or if a participant is presently receiving (or has received within 6 months prior to screening) anti-viral therapy for hepatitis C
* Clinically significant, active bacterial, viral, fungal, or parasitic infection (based on Investigator's judgement)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2030-04-02 (Estimated); Study Completion 2030-04-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline to Week 260

SECONDARY OUTCOMES:
Proportion of participants with sustained plasma level of Phe<360 μmol/L for ≥4 weeks without dietary Phe restriction at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Change from baseline in plasma level of Phe at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Change from baseline in dietary protein intake at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Proportion of participants with sustained plasma level of Phe <600 μmol/L for ≥ 4 weeks without dietary Phe restriction at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Proportion of participants with sustained plasma level of Phe <120 μmol/L for ≥ 4 weeks without dietary Phe restriction at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Change from baseline in plasma Phe: Tyr ratio at Week 24, 48, and Week 96 or Early Termination Visit following SAR444836 administration | From Baseline to Week 96
Number of participants with abnormal laboratory chemistry values | From Baseline to Week 96
Assessment of the duration of viral vector shedding of SAR444836 in sampling of urine, saliva, and semen at 4-week intervals following SAR444836 administration | From Baseline to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- United States (7):
  - University of California San Francisco- Site Number : 8400007, San Francisco, California
  - Children's Hospital IMD Clinic- Site Number : 8400015, Aurora, Colorado
  - University of Florida-Genetics- Site Number : 8400010, Gainesville, Florida
  - UHCMC- Site Number : 8400014, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh-4401 Penn Ave- Site Number : 8400018, Pittsburgh, Pennsylvania
  - Medical University of SC- Site Number : 8400004, Charleston, South Carolina
  - University of Texas- Site Number : 8400002, Houston, Texas
- Investigational Site Number : 0320002, Ciudad Autonoma Buenos Aires, Buenos Aires, Argentina
- Hospital de Clinicas de Porto Alegre - HCPA- Site Number : 0760001, Porto Alegre, Rio Grande do Sul, Brazil
- Investigational Site Number : 3760001, Tel Litwinsky, Israel
- Investigational Site Number : 7920001, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DFI17545 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25223&tenant=MT_SNY_9011